CLINICAL TRIAL: NCT06753188
Title: Clinical Pattern of Glanzemnn Thrombathenia in Children Attending Assiut University Children Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abeer Abd El Wahab Hassan Gomaa, resident doctor at Assiut University hospital, Assiut University
Other Study IDs: Glanzemnn thrombathenia AUCH
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Glanzemnn Thrombathenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- group 1: responder (complete sessation of bleeding) within 1-3 doses.
- group 2: partially responders who need more than 3 doses (3-5 dose for control of bleeding)
- group 3: non responder and need platelet concentarat transfusion Addationaly, duration of hospital stay, need for PRBC transfusion and ICU admission rate will be evaluated in all groups.

SUMMARY:
there are major limitations of these GTR data, they were not obtained using a defined treatment protocol in a randomized manner and treatment effectiveness and safety were not assessed at multiple, consistent, predefined time points. Furthermore, the frequent use of multiple agents in GT and delays in obtaining platelets make it particularly difficult to attribute effectiveness to any one or more products effectiveness and safety of using rFVII in pediatric cardiac surgery using data from existing double-arm studies.The administration of rFVII does not provide any added advantage forbleeding control among pediatric patients of cardiac surgery. However, it increased the rate of reexploration among the intervention arm Addationaly, Man-Chiu Poon et.al concluded that despite the results of GTR, there is a need for more data to support the efficacy and safety of rFVIIa in patients without platelet antibodies, without refractoriness to platelets and in cases when platelets are not readily available.

This study aimed to demonstrate the clinical pattern of Glanzemnn thrombathenia in children attending Assiut University Children Hospital

DETAILED DESCRIPTION:
Glanzmann's thrombasthenia, which is a rare autosomal recessive inherited platelet disorder characterised by impaired platelet aggregation and due to defects in the platelet membrane glycoprotein (GP) IIb-IIIa(1)With a prevalence of 1:1 million, GT is rare, although the prevalence is higher in areas where marriage between relatives is common(2 ,3 )The exact incidence has been difficult to calculate, but is estimated at one in 1,000,000. With an autosomal recessive inheritance, males and females are affected equally. There is a worldwide distribution; however, a large proportion of the cases have been described in selected populations such as the French Romani(16)South Indian Hindus, Iraqi Jews, and Jordanian nomadic tribes(17).Type I is the most common subtype and accounts for around 78% of patients with GT type II and type III (functional variant in receptor) constituting around 14% and 8% of cases (19) most patients present with severe mucocutaneous bleeding at an early age. A classic pattern of abnormal platelet aggregation, platelet glycoprotein expression and molecular studies confirm the diagnosis. Bleeding manifestations range from easy bruising, purpura, epistaxis, gingival bleeds, haematuria, haemarthrosis, muscle haematomas to central nervous system bleed.( 1 )Epistaxis is the most common cause of severe bleeding,risk of severe nosebleeds decreases with age as the septal arterial plexus becomes less friable and children grow out of the habit of nose picking,Menorrhagia is highly prevalent in affected females and there is a higher risk of severe bleeding at the time of menarche due to the prolonged estrogen influence on the proliferative endometrium that occurs during anovulatory cycles.Several bleeding scores have been developed with the goal of standardizing the assessment of bleeding and facilitating the diagnosis of patients with a suspected inherited bleeding disorder.(18) which usually appear in early childhood , among the 187 patients with a known age of onset of bleeding, 53% had bleeding symptoms by 1 year of age and 85% by 14 years of age (median and mean ages of onset were 1 year and 5.6 years, respectively). ( 1 , 4 ,5 )Management of bleeding is based on a combination of hemostatic agents including recombinant activated factor VII with or without platelet transfusions and antifibrinolytic agents. Platelet transfusion is the standard of care if the bleeding is unresponsive to these conservative means. (5 ,6) However, platelet transfusion has several limitations including potential for blood-borne pathogen transmission, particularly bacterial infection. (7 , 8 )Patients may develop antibodies to human leucocyte antigen (HLA) or integrin α2bβ3, which can lead to platelet refractoriness, making future transfusions ineffective. (5 , 6)platelets may not be readily available in emergencies(.4). rFVIIa is being increasingly used in certain disorders of platelet dysfunction, particularly Glanzmann's thrombasthenia(1)The haemostatic effect of pharmacological doses of rFVIIa seems to be that of enhancing the rate of thrombin generation on thrombin-activated platelet surfaces, thus providing the thrombin necessary for the formation of a stable fibrin haemostatic plug. Based on this information, rFVIIa has also been employed in disorders characterised by impaired thrombin generation, such as quantitative and qualitative platelet defects.Recombinant activated factor VII (rFVIIa; eptacog alfa activated, NovoSeven, Novo Nordisk A/S, Bagsværd, Denmark) was approved by the European Medicines Agency (EMA) in 2004 for the treatment of bleeding episodes and for the prevention of bleeding during surgery or invasive procedures in patients with GT.

The GT Registry (GTR) was an international, multicenter, observational registry that focused on both adults and children, aims to evaluate rFVIIa effectiveness and safety as a treatment for young patients with GT. The GTR was set up as a part of an EMA regulatory commitment to collect postmarketing data on rFVIIa utilization in patients with GT. Data on the use of other therapeutic options (platelets and antifibrinolytics) were also collected.

Data from GTR found that rFVIIa, provided effective hemostasis with a low frequency of adverse events in surgical, as well as nonsurgical, bleeding in patients with GT. The data from GTR support the applicability of rFVIIa as a good alternative treatment to platelet transfusions for severe bleeding episodes .

ELIGIBILITY:
Inclusion Criteria:

1. Age from one month to 18 year
2. Both sexes
3. Patients diagnosed to have Glanzemnn thrombathenia admitted with active bleeding.

Exclusion Criteria:

1. Patients less than one month and more than 18years
2. All other caused of congenital or acquired bleeding disorders in children including diseases treated with rFVII eg haemophilia with inhibitors

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed to have Glanzemnn thrombathenia admitted with active bleeding.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
response rate | 30 day
  response rate after patients will recived combine of rFVII Tranximic acid in adose of 10 mg/kg/dose IV /12 hour

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nurden AT, Fiore M, Nurden P, Pillois X. Glanzmann thrombasthenia: a review of ITGA2B and ITGB3 defects with emphasis on variants, phenotypic variability, and mouse models. Blood. 2011 Dec 1;118(23):5996-6005. doi: 10.1182/blood-2011-07-365635. Epub 2011 Sep 13. PMID 21917754
- [Background] Vamvakas EC, Blajchman MA. Blood still kills: six strategies to further reduce allogeneic blood transfusion-related mortality. Transfus Med Rev. 2010 Apr;24(2):77-124. doi: 10.1016/j.tmrv.2009.11.001. PMID 20303034
- [Background] Poon MC, d'Oiron R. Alloimmunization in Congenital Deficiencies of Platelet Surface Glycoproteins: Focus on Glanzmann's Thrombasthenia and Bernard-Soulier's Syndrome. Semin Thromb Hemost. 2018 Sep;44(6):604-614. doi: 10.1055/s-0038-1648233. Epub 2018 Jun 7. PMID 29879742
- [Background] Toogeh G, Sharifian R, Lak M, Safaee R, Artoni A, Peyvandi F. Presentation and pattern of symptoms in 382 patients with Glanzmann thrombasthenia in Iran. Am J Hematol. 2004 Oct;77(2):198-9. doi: 10.1002/ajh.20159. PMID 15389911